CLINICAL TRIAL: NCT01661426
Title: Weight Loss Diet Study: Low Carbohydrate vs. Low Fat and Insulin Resistance Status
Brief Title: Weight Loss Diet Study: Low Carb vs Low Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Associate Professor of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SU-07262012-10669
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Insulin Resistance
Keywords: Adults; Weight loss; Diet; Insulin Resistance; Fatty acid composition
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: The study employed a 2 x 2 crossover design: LF vs. LC diets and more IR vs. more IS. Study participants were classified as more IR or more IS based on the median AUC for insulin concentrations measured from an oral glucose tolerance test (OGTT) prior to randomization. Participants above the median were considered more IR and those below the median were considered more IS. A random number generator was used to stratify the randomization to LF vs. LC by insulin resistance status and gender. Participants followed their assigned diet for 6 months and then switched to the opposite diet for another 6 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Carbohydrate Diet first, then Low-Fat Diet (IR) (Active Comparator): Participants who were more insulin resistant based on the median AUC for insulin concentrations measured from OGTT prior to randomization.
  Interventions: Behavioral: Low-Carbohydrate Diet; Behavioral: Low-Fat Diet
- Low-Fat Diet first, then Low-Carbohydrate Diet (IS) (Active Comparator): Participants who were more insulin sensitive based on the median AUC for insulin concentrations measured from OGTT prior to randomization.
  Interventions: Behavioral: Low-Carbohydrate Diet; Behavioral: Low-Fat Diet

INTERVENTIONS:
Behavioral: Low-Carbohydrate Diet — Counseling/instruction on how to follow a healthy low-carbohydrate diet for 6 months. One evening class/week for 8 weeks (8 total classes). Then one class every other week for 8 weeks (4 total classes). Then one class every four weeks for 8 weeks (2 total classes): 14 evening classes, total.
Behavioral: Low-Fat Diet — Counseling/instruction on how to follow a healthy low-fat diet for 6 months. One evening class/week for 8 weeks (8 total classes). Then one class every other week for 8 weeks (4 total classes). Then one class every four weeks for 8 weeks (2 total classes): 14 evening classes, total.

SUMMARY:
The traditional weight loss diet recommended by health professionals has been a low-fat, high-carbohydrate, calorie restricted diet. This recommendation has been challenged by a number of alternative dietary strategies, particularly low-carbohydrate diets. In several recent weight loss studies insulin resistant adults had more success with low- vs. high-carbohydrate diets, in contrast to insulin sensitive adults who had either more success or comparable success with the low-fat diets. The investigators enrolled 61 people with a wide range of insulin sensitivity/resistance. After determining their insulin resistance status, the investigators will split them in the middle and randomly assign them to one of four groups for six months: (1) Low-Carbohydrate/Insulin Resistant (LC/IR); (2) Low-Carbohydrate/Insulin Sensitive (LC/IS); (3) Low-Fat/Insulin Resistant (LF/IR); and (4) Low-Fat/Insulin Sensitive (LF/IS) (15 people/group). After 6 months the participants will switch diet for the following 6 months, i.e. those randomized to the Low-Carbohydrate diet will switch to the Low-Fat diet and vice-versa. The primary outcome of this study is to determine whether weight loss success can be increased if one follows the dietary approach appropriately matched to their insulin resistance status. Secondary outcomes include fasting insulin, glucose, lipids, and fatty acid composition.

--------------------------------------------------------------------------------

DETAILED DESCRIPTION:
The investigators hope to learn whether matching the weight loss diet to one's insulin resistance status will increase weight loss the success. The relevance of these findings is highlighted by the fact that the national recommendations for weight loss are to follow a high-carbohydrate, low-fat diet. This would imply that about half the population has been given the wrong advice in regards to the most successful dietary pattern for weight loss.

Plasma fatty acid composition patterns have been shown to be associated with both insulin resistance and/or carbohydrate intake. As secondary analyses, the investigators will explore: (1) differences in plasma fatty acid composition between insulin sensitive and resistant participants at baseline; (2) the correlations between insulin markers and plasma fatty acid composition at baseline; (3) the interaction between insulin status and diet on 6-month changes in the plasma fatty acid composition; (4) plasma fatty acid composition changes in participants on low fat and low carbohydrate diets after 6 months; and (5) the correlations between changes in insulin markers, dietary components, and plasma fatty acid composition after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or = 18 years of age
* Women: Pre-menopausal (self-report) and <50 years of age
* Men: <50 years of age
* Race/Ethnicity: All
* BMI (body mass index): 28-40 kg/m2 (need to lose >10% body weight to achieve healthy BMI)
* Body weight stable for the last two months, and not actively on a weight loss plan
* No plans to move from the area over the next 14 months
* Available and able to participate in the evaluations and intervention for the study period
* Willing to accept random assignment
* To enhance study generalizability, people on medications not noted below as specific exclusions can participate if they have been stable on such medications for at least three months
* Ability and willingness to give written informed consent
* No known active psychiatric illness

Exclusion Criteria:

* Pregnant, lactating, within 6 months post-partum, or planning to become pregnant in the next 12 months; no menstruation for the previous 12 months
* Diabetes (type 1 and 2) or history of gestational diabetes or on hypoglycemic medications for any other indication
* Prevalent diseases: Malabsorption, renal or liver disease, active neoplasms, recent myocardial infarction, hypertension (except for those stable on hypertensive medications) (<6 months) (patient self-report and, if available, review of labs from primary care provider)
* Smokers (because of effect on weight and lipids)
* History of serious arrhythmias, or cerebrovascular disease
* Uncontrolled hyper- or hypothyroidism (TSH not within normal limits)
* Medications: Lipid lowering, diabetes medications, and those known to affect weight/energy expenditure
* Excessive alcohol intake (self-reported, >3 drinks/day)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline and 12 months
  Weight change was calculated as the 12 month value minus the baseline value

SECONDARY OUTCOMES:
Change in Fasting Insulin | Baseline and 12 months
  Fasting insulin change was calculated as the 12 month value minus the baseline value
Change in insulin AUC | Baseline and 12 months
  Insulin area under the curve (AUC) change was calculated as the 12 month value minus the baseline value.
Change in Fasting Glucose | Baseline and 12 months
  Fasting glucose change was calculated as the 12 month value minus the baseline value.
Change in LDL-Cholesterol | Baseline and 12 months
  LDL-cholesterol change was calculated as the 12 month value minus the baseline value.
Change in HDL-Cholesterol | Baseline and 12 months
  HDL-cholesterol change was calculated as the 12 month value minus the baseline value.
Change in Triglycerides | Baseline and 12 months
  Triglycerides change was calculated as the 12 month value minus the baseline value.
Change in systolic and diastolic blood pressure | Baseline and 12 months
  Blood pressure change was calculated as the 12 month value minus the baseline value.
Plasma fatty acid composition at baseline | Baseline
  Comparison of the plasma fatty acid composition between insulin sensitive and resistant participants at baseline.
Correlations between insulin markers and plasma fatty acid composition at baseline. | Baseline
Interaction between insulin status and diet on 6-month changes in the plasma fatty acid composition. | 6 months
Comparison of plasma fatty acid composition changes in participants on low fat and low carbohydrate diets after 6 months. | Baseline and 6 months
Correlations between changes in insulin markers, dietary components, and plasma fatty acid composition after 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardner CD, Offringa LC, Hartle JC, Kapphahn K, Cherin R. Weight loss on low-fat vs. low-carbohydrate diets by insulin resistance status among overweight adults and adults with obesity: A randomized pilot trial. Obesity (Silver Spring). 2016 Jan;24(1):79-86. doi: 10.1002/oby.21331. Epub 2015 Dec 6. PMID 26638192
- See also: Study description and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/different-diets-and-insulin-resistance.html